CLINICAL TRIAL: NCT06085963
Title: Nasal Allergen Challenge Test as a Method to Detect Clinical Reactivity Against Birch Pollen
Acronym: NAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars Olaf Cardell, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EudraCT: 2021-004632-29; K 2023-7697 (Other: Karolinska University Hospital)
Record Dates: First submitted 2023-09-27; First posted 2023-10-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Allergic Rhinitis Due to Pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 20 non-atopic controls will be randomized to dissolved placebo-tablet or saline solution in a cross over design. . This will be performed in a one side blinded challenge where 10 subjects will start with placebo-tablet dissolved in 0,9% saline solution and 10 will start with 0,9% saline solution only. After 30 minutes subjects will receive the other solution.
  Thereafter 70 patients will initially receive a NAC with 0,9% saline solution to ensure negative reactivity to the challenge as method. If negative after 30 minutes NAC will continue with one puff (1x0.1 ml) dissolved ITULAZAX® (1 SQ-Bet/ml) in each nostril.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 20 subjects will be challenged with both a dissolved placebo-tablet and 0.9% saline solution. This provocation will be performed as a one-sided blinded challenge which will demonstrate that the NAC is truly negative.
  Subjects will be randomized to dissolved placebo-tablet or saline solution in a cross over design. 10 subjects will start with dissolved placebo-tablet and 10 will start with 0.9% saline solution. After 30 minutes the subjects will switch to receive a challenge with the other solution. This will ensure negative reactivity to the excipients and challenge as a method. The placebo solution will be prepared the same as way as the active ITULAZAX® stock solutio
  Interventions: Drug: Placebo tablet; Drug: Nacl
- Birch group (Active Comparator): NAC will be applied to 70 patients with birch pollen allergy. Subjects will initially receive a NAC with 0,9% saline solution to ensure negative reactivity to the challenge as method. If negative after 30 minutes NAC will continue with one puff (1x0.1 ml) dissolved ITULAZAX® (1 SQ-Bet/ml) in each nostril.
  Interventions: Drug: ITULAZAX 12 SQ-Bet; Drug: Nacl

INTERVENTIONS:
Drug: ITULAZAX 12 SQ-Bet — Active ingredients: Birch (Betula verrucosa) extracts Dosage form: Oral lyophilisate (referred to as allergy immunotherapy tablet in text) Dose/strength: 12 SQ-Bet Excipients: Gelatine (fish source), mannitol and sodium hydroxide
  Arms: Birch group
Drug: Placebo tablet — Active ingredients: None Dosage form: Oral lyophilisate (referred to as allergy immunotherapy tablet in text) Excipients: Gelatine (fish source), mannitol and sodium hydroxide
  Arms: Control group
Drug: Nacl — Sodium chloride solution 9mg/ml

SUMMARY:
Clinical efficacy and tolerability for allergen specific immunotherapy (AIT) with Itulazax (birch pollen extract tablet) is well established.

Allergen challenges are used by clinicians to confirm correct diagnosis and by researchers to evaluate the efficacy of different interventions, eg. AIT. The challenge is performed by using a specific controlled administration schedule of an allergen product in the shock organ (nose, eye, or airway) and then monitor the result. Nasal Allergen Challenge (NAC) is the most common allergen challenge used.

Aquagen SQ (birch pollen extract) has since decades been golden standard for this purpose, but production of this product ended 2019. Clinicians as well as researchers are now in need for an alternative product.

To evaluate a new method for NAC would be of value from a clinical- and research perspective. From a Nordic perspective a NAC study with dissolved Itulazax would be of special interest since birch allergy is a dominant allergen in the region. In a recently published article it was shown that dissolved Grazax and Aquagen Phleum pratense gave comparable result used in grass allergic patients. Therefore, it seems reasonable to assume that the same method could be used with dissolved Itulazax.

The aim of this clinical trial is to evaluate the feasibility of nasal allergen challenge tests with dissolved Itulazax tablets. The main benefit of this proposal is that the allergen composition of the provocation test product is the same as the final product to be treated with. This is likely to increase the treatment motivation of the patient. In addition, the dissolving process is easier for the physician compared to the dissolving of the previously used Aquagen.

DETAILED DESCRIPTION:
The objective of the trial is to establish a method for Nasal Allergen Challenge (NAC) with dissolved Itulazax.

This trial is an open-label, national, one-centre trial comparing the results of NAC applied by solutions of dilutions of dissolved Itulazax tablets with the clinical diagnosis of birch pollen allergy by an experienced physician.

To ensure negative reactivity to the excipients of the tablet and the nasal provocation itself a non-atopic control group of 20 subjects will be challenged with both a dissolved placebo-tablet and 0.9% saline solution. This provocation will be performed as a one-sided blinded challenge which will demonstrate that the NAC is truly negative.

Thereafter 70 patients will initially receive a NAC with 0,9% saline solution to ensure negative reactivity to the challenge as method. If negative after 30 minutes NAC will continue with one puff (1x0.1 ml) dissolved Itulazax (1 SQ-Bet/ml) in each nostril. Total nasal symptom scores (TNSS, 0-12) and peak nasal inspiratory flow (PNIF) will be recorded before NAC and then at 5, 15 and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related assessments are performed
* Male or female aged 18-65 years at the time of consent
* A female subject of child-bearing potential must have a negative pregnancy test and be willing to practise appropriate highly effective birth control methods. The definition of a female patient of childbearing potential is a nonmenopausal female who has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure.
* The subject must be willing and able to comply with the trial protocol
* Birch pollen allergy group: A documented clinically relevant history of moderate to severe persistent birch pollen allergy symptoms since at least 2 years with troublesome symptoms despite the use of symptomatic medication with or without asthma; positive SPT(skin prick testing) response (wheal diameter ≥3 mm) to birch pollen (birch) and positive specific IgE (immunoglobulin E) to birch (≥ IgE CAP(quantitative test that measures the overall quantity of circulating IgE in the blood) class 2; ≥0.70 kU/L) at screening.
* Non-allergic control group: A documented negative clinical history for allergic rhinitis, negative SPT response (wheal diameter <3 mm) and negative sIgE (IgE CAP class 0) to birch pollen (birch), grasses, house dust mite, cat, horse, dog, ragweed, mugwort and mould (Alternaria alternata).

Exclusion Criteria:

* A subject in the birch pollen allergy group with rhinitis and/or conjunctivitis caused by animal hair and dander to which the subject is regularly exposed is not eligible for the trial. In terms of seasonal and perennial allergens like moulds etc. the subject can be sensitised to these allergens but is not eligible for the trial if the subject has symptoms induced by these allergens during the trial period.
* Patients who have experienced a severe asthma exacerbation within the last 3 months.
* Reduced lung function (in adults: FEV1 (Forced Expiratory Volume 1 sec) < 70% of predicted value after adequate pharmacologic treatment).
* SLIT (sublingual immunotherapy) treatment with birch pollen for more than 1 month within the last 5 years. In addition, any SLIT treatment with birch pollen within the previous 12 months.
* SCIT (subcutaneous immunotherapy) treatment with birch pollen reaching the maintenance dose within the last 5 years. In addition, any SCIT treatment with birch pollen within the previous 12 months.
* Ongoing treatment with any allergy immunotherapy product
* Has any nasal oropharyngeal condition that might mimic birch pollen allergy symptoms (e.g. strong septal deviation, nasal polyps, a history of paranasal sinus surgery or surgery of nasal turbinate's; choanal atresia, hypertrophy of pharyngeal tonsil, naso/oropharyngeal tumours, hypertrophy of palatial tonsils). For exclusion both sided nasal endoscopy including endoscopy of the epipharynx is required.
* Any general condition that might induce birch pollen allergy symptoms (hypothyroidism, pregnancy).
* Any pharmacotherapy that might induce birch pollen symptoms (e.g. treatment with antihypertensive drugs, treatment with cholinergic acting drugs like antidepressants).
* History of any other (allergic) rhinitis symptoms than to birch pollen during the whole study period for subjects in the birch pollen allergy group.
* A relevant history of systemic allergic reaction e.g. anaphylaxis with cardiorespiratory symptoms, generalised urticaria or severe facial angioedema that in the opinion of the investigator may constitute an increased safety concern.
* Any clinically relevant chronic disease incl. malignancy that in the opinion of the investigator would interfere with the trial evaluations or the safety of the subject.
* Active or poorly controlled autoimmune diseases, immune defects, immunodeficiencies, immunosuppression or malignant neoplastic diseases with current disease relevance.
* Immunosuppressive treatment (ATC code L04 or L01) within 3 months prior to the screening visit.

  ·-Treatment with medications with potential impact on NAC (e.g. treatment with anti-IgE or anti IL-5 (interleukin 5) drugs within 130 days/5 half-lives of the drug (which ever longest) or treatment with antidepressant or antipsychotic medications with antihistaminic effect).
* Current participation in other clinical trials and or use of an investigational drug within 30 days/5 half-lives of the drug, which ever the longest, prior to screening.
* A history of allergy, hypersensitivity or intolerance to the IMP (investigation medicinal product) (except birch pollen).
* Smoking / significant history of smoking.
* A history of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
TNSS | The symptoms are scored 5,15 and 30 minutes after provocation
  0,1 x ml of dissolved Itulazax or NaCl will be sprayed into each nostril. The change from baseline (TNSS before provocation) in Total Nasal Symptom Score (TNSS) will be measured 5,15 and 30 minutes after negative (NaCl) and positive provocation (Itulazax). Subjective measures will be made by a Total Nasal Symptom Score (TNSS) on a 0-12 Likert scale. Increase of ≥5 points indicates clearly positive test. Increase of ≥3 points indicates moderately positive test
PNIF | The symptoms are scored 5,15 and 30 minutes after provocation.
  0,1 x ml of dissolved Itulazax or NaCl will be sprayed into each nostril. Peak nasal inspiratory flow (PNIF) wil be meaused with a PNIF Meter. The change from baseline (PNIF before provocation) in Peak Nasal Inspiratory Flow (PNIF) will be measured 5,15 and 30 minutes after negative (NaCl) and positive provocation (Itulazax). Objective measures will be an assessment of the Peak Nasal Inspiratory Flow (PNIF). Flow decrease of ≥40% indicates clearly positive test. Flow decrease of ≥20% indicates moderately positive test.

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olaf Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No